CLINICAL TRIAL: NCT02588274
Title: Efficacy of Acupuncture for Chronic Prostatitis/Chronic Pelvic Pain Syndrome: Study Protocol for a Randomized, Placebo-controlled Trial
Brief Title: Efficacy of Acupuncture for Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Qin Zongshi, Doctor of Department of Acupuncture, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015S102
Record Dates: First submitted 2015-10-20; First posted 2015-10-27 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Chronic Prostatitis
Keywords: Chronic prostatitis; chronic pelvic pain syndrome; acupuncture; placebo needle; randomized controlled trial
MeSH Terms: interventions — Acupuncture Therapy; Needles

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Zhongliao (BL 33), Shenshu (BL 23), Huiyang (BL 35), and Sanyinjiao (SP 6) acupuncture points (Table 1). After patients are in prone position with relax, the investigators will use 75% alcohol pads to sterile the skin around the acupuncture points, and then insert steel needles (Huatuo, Suzhou, China 0.3mm*40mm/0.3mm*75mm) into the acupuncture points. For bilateral Zhongliao (BL 33), the needle will be inserted into about 50-60mm with 45 degree, for Huiyang (BL 35), the needle will be inserted into 50-60mm. for Shenshu (BL 23) and Sanyinjiao (SP 6), the needles will be inserted vertically to a depth of 25-30 mm. The treatment sessions are 24 after baseline, 3 times a week, and the each time the patients will accept a 30 minutes treatment.
  Interventions: Device: Acupuncture
- placebo needle (Placebo Comparator): The participants in placebo needle group will receive placebo needle at the same acupuncture points to treatment group. Investigators will use a sort of blunt needle that cannot penetrate skin and stimulate deep tissues while the thrusting and twisting manipulation will be used by acupuncturists to mock the treatment procedure and blind the patients. The duration and frequency of sessions are same to the treatment group.
  Interventions: Device: placebo needle

INTERVENTIONS:
Device: Acupuncture — Acupuncture is one of the oldest standardized neuromodulatory therapies. The method of acupuncture treatment involves the insertion of needles in acupuncture points according to a system of channels and meridians. The needles are stimulated by manual manipulation, electrical stimulation or heat. The general theory of acupuncture is based on the premise that there are patterns of energy flow through the body that are essential for health. Disruptions of this flow are believed to be responsible for disease. Acupuncture may correct imbalances of flow at identifiable points close to the skin.
  Other Names: needle
  Arms: Acupuncture
Device: placebo needle — Placebo needle is a type of control without skin penetration based on the application of placebo needles with blunt needle tips.
  Arms: placebo needle

SUMMARY:
Chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) affects many adult men worldwide. So far, available therapies offer little or no proven benefit to CP/CPPS. The investigators design and implement this study is to assess efficacy of acupuncture therapy performed in the CP/CPPS .

DETAILED DESCRIPTION:
This study is a multi-center, placebo-controlled, randomized trial comparing acupuncture and placebo needle among patients with CP/CPPS, which will be conducted in Guang'anmen Hospital of China Academy of Chinese Medical Sciences and Yantai Chinese Medicine Hospital from November 2015 to May 2017. 68 patients will be recruited in total through the advertisements spreading by newspaper, television and internet. After participants have completed a baseline evaluation and meet the selection criteria, one professional statistician uninvolved with treatment and data collection will assigns the participants by using a computer generated, blocked random allocation sequence randomly and acupuncturist will be blinded to the process of randomized assignment.Treatment group will use acupuncture and control group will use placebo needle, for treatment, Zhongliao (BL 33), Shenshu (BL 23), Guiyang (BL 35), Sanyinjiao (SP 6) acupuncture points will be used, the treatment sessions are 24 weeks after baseline, 3 times a week and each time the patients will accept a 30 minutes treatment, to control group, participants will receive placebo needle treatment at the same acupuncture points and the duration and frequency of sessions are same to the real acupuncture group. The primary outcome measure of this study is the decreasing in (National Institutes of Health Chronic Prostatitis Symptom Index) NIH-CPSI total score from baseline to week 8, and secondary outcomes include NIH-CPSI sub scales at week, (International Prostate Symptom Score) IPSS total score, Global response assessment, expectation degree and satisfaction degree. The first three secondary outcomes will be measured at 4,8,20 and 32 weeks, expectation degree will be measured at baseline, and the satisfaction degree will be measure at 8, 20, 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. History of pain perceived in the region of the prostate and absence of other lower urinary tract pathology for a minimum of 3 out of the past 6 months. In addition, associated lower urinary tract symptoms, sexual function, psychological factors should be addressed.
2. Age 18 to 50 years
3. NIH Chronic Prostatitis Symptom Index (NIH-CPSI) total score≥ 15 (scale 0-43, and 0 means no symptom).

Exclusion Criteria:

1. Other urologic disease (for example, acute prostatitis, bacterial prostatitis, benign prostatic hyperplasia, prostate cancer, urinary tuberculosis, urinary tract infection)
2. Serious or acute diseases with heart, liver, kidney and blood system.
3. Patients who had received acupuncture or medication (including alpha-blockers or pain killers) treatment in the week prior to the baseline assessment
4. Patients without telephone number who cannot be connected during the follow-up

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
NIH-CPSI total score and change from baseline | baseline, week 1-8

SECONDARY OUTCOMES:
NIH-CPSI subscales score | Baseline, week 4,8,20,32
NIH-CPSI total score in follow-up | week 20,32
IPSS total score and change from baseline | baseline, week 4,8,20,32
Global response assessment improvement | week 4,8,20,32
expectations degree | baseline
  The expectations that acupuncture might help participants CP/CPPS at baseline. This scale includes two brief questions to investigate whether patients believe acupuncture treatment and if acupuncture may help CP/CPPS. The investigators designed this scale and the investigators want to explore the impact of variable that are potentially associated with placebo effects, namely will participants' expectations be treatment effect modifier?
Degree of satisfaction | week 8,20,32
  The investigators designed this scale, which include 5 grades answer from 0 to 4, means "not at all" "a little" "Quite satisfied" "satisfaction" "very satisfaction"and the investigators want to use this to test blinding of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, PhD, Principal Investigator — Guang'anmen Hospital
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Science, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Qin Z, Zang Z, Wu J, Zhou J, Liu Z. Efficacy of acupuncture for chronic prostatitis/chronic pelvic pain syndromes: study protocol for a randomized, sham acupuncture-controlled trial. BMC Complement Altern Med. 2016 Nov 7;16(1):440. doi: 10.1186/s12906-016-1428-y. PMID 27821109